CLINICAL TRIAL: NCT00375258
Title: A Large Randomised Placebo Controlled Trial Among Trauma Patients With, or at Risk of, Significant Haemorrhage, of the Effects of Antifibrinolytic Treatment on Death and Transfusion Requirement
Brief Title: Clinical Randomisation of an Antifibrinolytic in Significant Haemorrhage
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Professor Ian Roberts (Chief Investigator), London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISRCTN86750102
Record Dates: First submitted 2006-09-11; First posted 2006-09-12 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2011-06

CONDITIONS: Hemorrhage
Keywords: Adult trauma patients with ongoing significant haemorrhage or at risk of significant haemorrhage
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Active
  Interventions: Drug: Tranexamic acid
- 2 (Placebo Comparator)
  Interventions: Drug: Sodium Chloride 0.9%

INTERVENTIONS:
Drug: Tranexamic acid — Loading dose of 1 gram then 1 gram by infusion over 8 hours
  Arms: 1
Drug: Sodium Chloride 0.9% — Visual matched placebo
  Arms: 2

SUMMARY:
CRASH 2 is a large pragmatic randomised placebo controlled trial of the effects of the early administration of the antifibrinolytic agent tranexamic acid on death, vascular events and transfusion requirements. Adults with trauma who are within 8 hours of injury and have either significant haemorrhage, or who are considered to be at risk of significant haemorrhage, are eligible if the responsible doctor is for any reason substantially uncertain whether or not to use an antifibrinolytic agent. Numbered drug or placebo packs will be available in each participating emergency department. Randomisation will involve calling a 24-hour freecall randomisation service. The call should last only a minute or two and at the end of it the randomisation service will specify which numbered treatment pack to use. For hospitals where telephone randomisation is not feasible, randomisation will be by taking the next consecutively numbered treatment pack. No extra tests are required but a short form must be completed one month later or on discharge or on death (whichever occurs first).

DETAILED DESCRIPTION:
See trial website for full protocol. This is an international trial with over 300 hospitals in about 40 countries worldwide.

ELIGIBILITY:
Inclusion Criteria:

All trauma patients with ongoing significant haemorrhage (systolic blood pressure less than 90 mmHg and/or heart rate more than 110 beats per minute), or who are considered to be at risk of significant haemorrhage, and are within 8 hours of the injury, are eligible for trial entry if they appear to be at least 16 years old. Although entry is allowed up to 8 hours from injury, the earlier that patients can be treated the better.

Exclusion Criteria:

The fundamental eligibility criterion is the responsible doctor's 'uncertainty' as to whether or not to use an antifibrinolytic agent in a particular adult with traumatic haemorrhage. Patients for whom the responsible doctor considers there is a clear indication for antifibrinolytic therapy should not be randomised. Likewise, patients for whom there is considered to be a clear contraindication to antifibrinolytic therapy (such as, perhaps, those who have clinical evidence of a thrombotic disseminated intravascular coagulation) should not be randomised. Where the responsible doctor is substantially uncertain as to whether or not to use an antifibrinolytic, all these patients are eligible for randomisation and should be considered for the trial. There are no other pre-specified exclusion criteria

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20211 (Actual)
Dates: Start 2005-05; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Death in hospital within four weeks of injury (causes of death will be described to assess whether deaths were due to haemorrhage or vascular occlusion). | Death, discharge or four weeks post randomisation whichever occurs first.

SECONDARY OUTCOMES:
Receipt of a blood products transfusion, the number of units of blood products transfused, surgical intervention, and the occurrence of thrombo-embolic episodes | Death, discharge or four weeks post randomisation whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Roberts, MD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Over 50 countries Worldwide, London, United Kingdom

REFERENCES:
- [Background] Coats T, Hunt B, Roberts I, Shakur H. Antifibrinolytic agents in traumatic haemorrhage. PLoS Med. 2005 Mar;2(3):e64. doi: 10.1371/journal.pmed.0020064. Epub 2005 Mar 29. PMID 15783255
- [Derived] Edgar K, Roberts I, Sharples L. Including random centre effects in design, analysis and presentation of multi-centre trials. Trials. 2021 May 22;22(1):357. doi: 10.1186/s13063-021-05266-w. PMID 34022937
- [Derived] Kolin DA, Shakur-Still H, Bello A, Chaudhri R, Bates I, Roberts I. Risk factors for blood transfusion in traumatic and postpartum hemorrhage patients: Analysis of the CRASH-2 and WOMAN trials. PLoS One. 2020 Jun 3;15(6):e0233274. doi: 10.1371/journal.pone.0233274. eCollection 2020. PMID 32492040
- [Derived] Nishijima DK, Kuppermann N, Roberts I, VanBuren JM, Tancredi DJ. The Effect of Tranexamic Acid on Functional Outcomes: An Exploratory Analysis of the CRASH-2 Randomized Controlled Trial. Ann Emerg Med. 2019 Jul;74(1):79-87. doi: 10.1016/j.annemergmed.2018.11.018. Epub 2019 Jan 12. PMID 30642657
- [Derived] Roberts I, Edwards P, Prieto D, Joshi M, Mahmood A, Ker K, Shakur H. Tranexamic acid in bleeding trauma patients: an exploration of benefits and harms. Trials. 2017 Jan 31;18(1):48. doi: 10.1186/s13063-016-1750-1. PMID 28143564
- [Derived] Roberts I, Prieto-Merino D, Manno D. Mechanism of action of tranexamic acid in bleeding trauma patients: an exploratory analysis of data from the CRASH-2 trial. Crit Care. 2014 Dec 13;18(6):685. doi: 10.1186/s13054-014-0685-8. PMID 25498484
- [Derived] Meurer WJ. Tranexamic acid reduced mortality in trauma patients who were bleeding or at risk for bleeding. Ann Intern Med. 2013 Sep 17;159(6):JC3. doi: 10.7326/0003-4819-159-6-201309170-02003. No abstract available. PMID 24042386
- [Derived] Roberts I, Shakur H, Coats T, Hunt B, Balogun E, Barnetson L, Cook L, Kawahara T, Perel P, Prieto-Merino D, Ramos M, Cairns J, Guerriero C. The CRASH-2 trial: a randomised controlled trial and economic evaluation of the effects of tranexamic acid on death, vascular occlusive events and transfusion requirement in bleeding trauma patients. Health Technol Assess. 2013 Mar;17(10):1-79. doi: 10.3310/hta17100. PMID 23477634
- [Derived] Williams-Johnson JA, McDonald AH, Strachan GG, Williams EW. Effects of tranexamic acid on death, vascular occlusive events, and blood transfusion in trauma patients with significant haemorrhage (CRASH-2) A randomised, placebo-controlled trial. West Indian Med J. 2010 Dec;59(6):612-24. PMID 21702233
- [Derived] Guerriero C, Cairns J, Perel P, Shakur H, Roberts I; CRASH 2 trial collaborators. Cost-effectiveness analysis of administering tranexamic acid to bleeding trauma patients using evidence from the CRASH-2 trial. PLoS One. 2011 May 3;6(5):e18987. doi: 10.1371/journal.pone.0018987. PMID 21559279
- [Derived] CRASH-2 collaborators; Roberts I, Shakur H, Afolabi A, Brohi K, Coats T, Dewan Y, Gando S, Guyatt G, Hunt BJ, Morales C, Perel P, Prieto-Merino D, Woolley T. The importance of early treatment with tranexamic acid in bleeding trauma patients: an exploratory analysis of the CRASH-2 randomised controlled trial. Lancet. 2011 Mar 26;377(9771):1096-101, 1101.e1-2. doi: 10.1016/S0140-6736(11)60278-X. PMID 21439633
- [Derived] CRASH-2 trial collaborators; Shakur H, Roberts I, Bautista R, Caballero J, Coats T, Dewan Y, El-Sayed H, Gogichaishvili T, Gupta S, Herrera J, Hunt B, Iribhogbe P, Izurieta M, Khamis H, Komolafe E, Marrero MA, Mejia-Mantilla J, Miranda J, Morales C, Olaomi O, Olldashi F, Perel P, Peto R, Ramana PV, Ravi RR, Yutthakasemsunt S. Effects of tranexamic acid on death, vascular occlusive events, and blood transfusion in trauma patients with significant haemorrhage (CRASH-2): a randomised, placebo-controlled trial. Lancet. 2010 Jul 3;376(9734):23-32. doi: 10.1016/S0140-6736(10)60835-5. Epub 2010 Jun 14. PMID 20554319
- See also: Trial website — http://www.crash2.lshtm.ac.uk